CLINICAL TRIAL: NCT07312773
Title: A Two-arm, Open-label, Single-sequence, Multiple-dose Study to Evaluate the Pharmacokinetic Interaction and the Safety of AD-231A and AD-231B and AD-231C in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetic Interaction and the Safety of AD-231A and AD-231B and AD-231C
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AD-231DDI
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Period 1 : Treatment A(AD-231A), Period 2 : Treatment C(AD-231A+AD-231B+AD-231C)
  Interventions: Drug: Treatment A(AD-231A); Drug: Treatment C(AD-231A+AD-231B+AD-231C)
- Arm B (Experimental): Period 1 : Treatment B(AD-231B+AD-231C), Period 2 : Treatment C(AD-231A+AD-231B+AD-231C)
  Interventions: Drug: Treatment B(AD-231B+AD-231C); Drug: Treatment C(AD-231A+AD-231B+AD-231C)

INTERVENTIONS:
Drug: Treatment A(AD-231A) — AD-231A Oral Tablet
  Arms: Arm A
Drug: Treatment B(AD-231B+AD-231C) — AD-231B+AD-231C Oral Tablet
  Arms: Arm B
Drug: Treatment C(AD-231A+AD-231B+AD-231C) — AD-231A+AD-231B+AD-231C Oral Tablet

SUMMARY:
To evaluate the pharmacokinetic interactions of AD-231A, AD-231B, and AD-231C in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged ≥19 and <65 years at the time of the screening visit
* Body weight ≥50 kg (≥45 kg for females) and body mass index (BMI) between 18.0 kg/m² and 30.0 kg/m² at the time of the screening visit

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve during dosing interval at steady state (AUCτ,ss) | pre-dose (0hour) to 24 hours post-dose on Day 14
  AUCτ,ss
Maximum concentration of drug in plasma at steady state (Cmax,ss) | pre-dose (0hour) to 24 hours post-dose on Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No